CLINICAL TRIAL: NCT07142356
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group, Multicenter Study of Modified Release RTN-001 In Patients With Uncontrolled Hypertension
Brief Title: A Study of Modified Release RTN-001 In Patients With Uncontrolled Hypertension
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Retension Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RTN-001-025-012
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Uncontrolled Hypertension
Keywords: hypertension; uncontrolled hypertension; RTN-001; blood pressure; systolic; diastolic
MeSH Terms: conditions — Hypertension; Systolic Murmurs; Heart Murmurs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RTN-001 (Experimental): RTN-001 will be administered orally. RTN-001 tablets will be provided in one dose strength (15 mg). Each patient will take 3 tablets daily of RTN-001, placebo, or both depending on assigned treatment group.
  Interventions: Drug: RTN-001
- Matching Placebo (Placebo Comparator): The reference/comparator product is a matching placebo tablet with similar appearance and weight as the RTN-001 oral tablet.
  Interventions: Drug: Matching placebo control

INTERVENTIONS:
Drug: RTN-001 — A potent and selective PDE5 inhibitor.
  Other Names: SLx-2101
  Arms: RTN-001
Drug: Matching placebo control — The reference/comparator product is a matching placebo tablet with similar appearance and weight as the RTN-001 oral tablet.
  Other Names: Placebo
  Arms: Matching Placebo

SUMMARY:
The goal of this clinical trial is to learn if the drug RT-001 works to reduce high blood pressure (hypertension) in adults. It will also learn about the safety of RTN-001. The main questions it aims to answer are:

Does RTN-001 lower blood pressure in patients who have uncontrolled hypertension? What medical problems do participants have when taking RTN-001?

Researchers will compare RTN-001 to a placebo (a look-alike substance that contains no drug) to see if RTN-001 works to treat uncontrolled hypertension.

Participants will:

Take RTN-001 or a placebo every day for 12 weeks Visit the clinic about once every 2 weeks for checkups and tests Keep a diary of their symptoms and all medications that they take including RTN-001

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, double-blind, parallel group, multicenter study conducted in the United States. Patients who have uncontrolled hypertension (SBP ≥ 130 mm Hg and DBP ≥ 80 mm Hg on ≥ 2 antihypertensive medications) and are aged 18 to 70 years, inclusive, will be eligible for screening. Patients will be stratified by the number of antihypertensive medications they are receiving (2 or ≥ 3), by sex (male, female), and by race (Black, non-Black).

The study consists of 3 periods, a Screening Period, a Run-in Period, and a Treatment Period. An Off-treatment (OT) Follow-up Visit will occur 2 weeks after conclusion of the Treatment Period.

The Screening Period (Visit S1) is up to 14 days in length (Days -28 to -15) and should occur no more than 28 days (± 7 days) before the randomization visit (Visit T1 [Day 1]). Patients who successfully complete all screening assessments at Visit S1 move on to the 14-day Run-in Period, which begins with Visit S2 (Day 14). The Run-in Period is single-blind (patients are blinded to the treatment they receive) to assess patient compliance with study drug and the patient's ability to undergo 24-hour ambulatory BP measurement. At Visit S2, patients will have peripheral (seated automated office BP measurement) and central BP measurements and be fitted with the monitor for their baseline 24-hour ambulatory BP measurement (ABPM). Successful completion of the Run-in Period requires > 80% dosing compliance and confirmation of valid data from baseline 24-hour ambulatory BP monitoring.

At the conclusion of the Run-in Period, approximately 280 eligible patients will enter the 12-week Treatment Period and be randomly assigned (1:1:1:1) to receive 12 weeks of QD treatment with RTN-001 at doses of 15, 30, or 45 mg or matching placebo.

On the morning of Visit T1 (Day 1), before the first administration of study drug, randomized patients will undergo baseline peripheral and central BP measurements and laboratory testing.

Patients will return for study visits at Week 2 (Visit T2 /Day 15), Week 4 (Visit T3/Day 29), Week 8 (Visit T4/Day 57), and Week 12 (Visit T5/Day 85/End of Study).

At each of the last 3 study site visits during the Treatment Period (Visits T3, T4, and T5), patients will undergo peripheral and central BP measurements. At these visits, as well as at Visit T2, patients will undergo blood sampling. Blood samples may be used for safety assessments, determination of drug and metabolite levels, and potential biomarker assessments. Ambulatory BP measurements will be obtained outside of the study site in the temporal proximity of the Week 4 and Week 12 study visit timepoints. A safety review may be conducted after approximately 25% of patients have completed the Week 2 (Visit T2) assessment. If no safety concerns are identified, the sponsor may choose to eliminate this visit from the study schedule.

Patients will receive an OT phone call on Day 99 (Visit OT) approximately 2 weeks after the last dose of RTN-001 or placebo to assess occurrence of adverse events and record changes in concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent before any study-specific procedure.
2. Male or female patients age 18 to 70 years, inclusive, at the Screening Visit.
3. Uncontrolled HTN despite being on a stable regimen of ≥ 2 antihypertensive medications in the following drug classes: ACE-inhibitors, ARBs, beta blockers, calcium channel blockers, mineralocorticoid receptor antagonists, or diuretics. A stable regimen is defined as being on the same medications and the same dose for at least 30 days before screening. A combination pill containing 2 separate classes of antihypertensive drugs is considered 2 antihypertensive medications.
4. Mean BP of ≥ 130/80 mm Hga.
5. Men and nonpregnant, nonlactating women. Women must be either:

   * Naturally postmenopausal defined as ≥ 1 year without menses and follicle-stimulating hormone ≥ 40.0 IU/L, or
   * Surgically sterile including hysterectomy, bilateral oophorectomy, and/or tubal ligation, or

   Women of childbearing potential must be willing to use 2 acceptable methods of birth control (unless they have agreed to follow the definition of true abstinence). The minimal requirement for adequate contraception should be started the day of Visit T1 (Day 1), continuing during the Treatment Period and for at least 30 days after the last dose of study drug. Acceptable methods of birth control include:
   * Oral, implantable, injectable, or topical birth control medications. Note: Oral birth control medication must be started ≥ 30 days before the first dose of treatment in the Placebo Run-in.
   * Placement of an intrauterine device with or without hormones.
   * Barrier methods including condom or occlusive cap with spermicidal foam or spermicidal jelly.
   * Vasectomized male partner who is the sole partner for this patient.
   * True abstinence when this is the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception.
6. Body mass index of 18 to 35 kg/m2.
7. Negative prestudy urine drugs of abuse screen (with the exception of tetrahydrocannabinol [THC]).
8. If taking a PDE5 inhibitor for erectile dysfunction, must be willing to pause use during the study period.

Only patients with uncontrolled HTN on ≥ 2 accepted classes of antihypertensive drugs who continue to satisfy the inclusion criteria above, are > 80% compliant during the Placebo Run-in dosing of 3 tablets QD of single-blind placebo and have successfully completed the baseline 24 hour ABPM will be randomly assigned to treatment with RTN-001 or matching placebo.

aThe initial BP inclusion criterion will be ≥ 130/80 mm Hg. After approximately 25% of patients (80 patients) have been randomly assigned to study treatment, the actual baseline BP of randomized patients will be reviewed to ensure target distribution of BP at study entry. If the mean baseline SBP is not within the target range of approximately 145 mm Hg, the inclusion criterion may be modified to reflect a higher BP inclusion criterion.

Exclusion Criteria:

1. Currently enrolled in a study with an investigational product or any other type of medical research within 30 days before randomization.
2. Mean seated SBP > 170 mm Hg and/or DBP > 110 mm Hg.
3. Current or planned use of nitrates and/or alpha-blockers or other drugs known to affect BP during the study period (except for those allowed in the protocol; Section 5.9.2) including SGLT2 inhibitors and GLP-1 agonists.
4. Regular user of PDE5 inhibitors or cannot/is unwilling to refrain from use of PDE5 inhibitors for 7 days before and during their participation in the study.
5. History of hypotension, fainting spells, or blackouts, including orthostatic hypotension.
6. Malignant HTN, primary aldosteronism, or secondary HTN.
7. Active pancreatitis.
8. A history of drug abuse.
9. Abuses alcohol defined as average weekly intake greater than 21 units for males or 14 units for females. One unit is equivalent to a 12 oz beer, 1 measure of spirits, or 1 glass of wine.
10. History or presence of gastrointestinal, hepatic, or renal disease or other conditions that would be known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
11. Recent (within 3 months before the Screening Visit [Visit S1]) myocardial infarction; unstable angina leading to hospitalization; uncontrolled, symptomatic cardiac arrhythmia (or medication for an arrhythmia that was started or dose changed within 3 months of screening); coronary artery bypass graft; percutaneous coronary intervention; carotid surgery or stenting; cerebrovascular accident; transient ischemic attack; endovascular procedure or surgical intervention for peripheral vascular disease; or plans to undergo a major surgical or interventional procedure (eg, percutaneous coronary intervention, coronary artery bypass graft, carotid or peripheral revascularization). Patients with implantable pacemakers or automatic implantable cardioverter defibrillators may be considered if deemed by the Investigator to be stable for the previous 3 months.
12. Uncontrolled hypothyroidism, including thyroid-stimulating hormone > 1.5 × the upper limit of normal (ULN) at the Screening Visit (Visit S1); patients stabilized on thyroid replacement therapy for at least 6 weeks before randomization are allowed.
13. Liver disease or dysfunction, including:

    1. Positive serology for hepatitis B surface antigen and/or hepatitis C antibodies at the Screening Visit (Visit S1), or
    2. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≥ 2 × ULN, and/or total bilirubin (TB) ≥ 2 × ULN at the Screening Visit (Visit S1). If TB ≥ 1.2 × ULN, a reflex indirect (unconjugated) bilirubin will be obtained, and if consistent with Gilbert's syndrome or if the patient has a history of Gilbert's syndrome, the patient may be enrolled in the study.

    Note: At the discretion of the Investigator, a repeat of ALT and/or AST may be completed before randomization. For those patients who have a repeat ALT and/or AST, the repeat value will be used to determine eligibility. Also, if the patient tests positive for the hepatitis C antibody, but the optional reflexive test for hepatitis C RNA is negative, the patient can be enrolled.
14. Renal dysfunction or glomerulonephritis, including estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) formula < 45 mL/min/1.73 m2 at the Screening Visit (Visit S1). Note: a single repeat qualifying eGFR, performed at the discretion of the Investigator, is acceptable.
15. Gastrointestinal conditions or procedures (including weight loss surgery [eg, Lap-Band or gastric bypass] that may affect drug absorption.
16. Hematologic or coagulation disorders or a hemoglobin level < 10.0 g/dL at the Screening Visit (Visit S1).
17. Active malignancy, including a malignancy requiring surgery, chemotherapy, and/or radiation in the 5 years before Screening. Nonmetastatic basal or squamous cell carcinoma of the skin and cervical carcinoma in situ are allowed.
18. Unexplained creatine kinase (CK) > 3 × ULN at any time before randomization, which is not associated with recent trauma or physically strenuous activity. Patients with an explained CK elevation must have a single repeat CK ≤ 3 × ULN before randomization.
19. Blood donation, participation in multiple blood draws, clinical study, major trauma, blood transfusion, or surgery with or without blood loss within 30 days before randomization.
20. Use of any experimental or investigational drug(s) within 30 days before Screening.
21. An employee or contractor of the facility conducting the study, or a family member of the principal investigator, co-investigator, or any Sponsor personnel
22. Is considered to be unsuitable for any other reason that may either place the patient at increased risk during participation or interfere with the interpretation of study outcomes by the Investigator, after reviewing the medical and psychiatric history, physical examination, and laboratory evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Mean change in systolic blood pressure at 4 weeks | 4 weeks
  The difference in the mean change in pre-dose office-seated systolic blood pressure in patients with uncontrolled hypertension after 4 weeks of treatment with RTN-001 versus placebo.

SECONDARY OUTCOMES:
Mean change in daytime ambulatory SBP at 4 weeks | 4 weeks
  Difference in mean change in daytime ambulatory SBP in patients with uncontrolled hypertension after 4 weeks of treatment with RTN-001 versus placebo.
Mean change in daytime ambulatory SBP at 8 and 12 weeks | 8 and 12 weeks
  Difference in the mean change in predose office-seated SBP in patients with uncontrolled hypertension after 8 and 12 weeks of treatment with RTN-001 versus placebo.
Mean change in pre-dose central SBP at 4 and 12 weeks | 4 and 12 weeks
  Difference in the mean change in predose central SBP in patients with uncontrolled hypertension after 4 and 12 weeks of treatment with RTN-001 versus placebo.
Mean change in daytime ambulatory SBP at 12 weeks | 12 weeks
  Difference in the mean change in daytime ambulatory SBP in patients with uncontrolled hypertension after 12 weeks of treatment with RTN-001 versus placebo.
Mean change in 24-hour ambulatory SBP at 4 and 12 weeks | 4 and 12 weeks
  Difference in the mean change in 24-hour ambulatory SBP in patients with uncontrolled hypertension after 4 and 12 weeks of treatment with RTN-001 versus placebo.
Mean change in predose office-seated DBP at 4, 8, and 12 weeks | 4, 8, and 12 weeks
  Difference in the mean change in predose office-seated DBP in patients with uncontrolled hypertension after 4, 8, and 12 weeks of treatment with RTN 001 versus placebo.
Mean change in predose central DBP at 4 and 12 weeks | 4 and 12 weeks
  Difference in the mean change in predose central DBP in patients with uncontrolled hypertension after 4 and 12 weeks of treatment with RTN-001 versus placebo.
Mean change in daytime ambulatory and 24-hour mean ambulatory DBP at 4 and 12 weeks | 4 and 12 weeks
  Difference in the mean change in daytime ambulatory and 24-hour mean ambulatory DBP in patients with uncontrolled hypertension after 4 and 12 weeks of treatment with RTN-001 versus placebo.
Percentage of patients achieving peripheral SBP < 130 mm Hg and/or DBP < 80 mm Hg at t=0 (predose) at 4, 8, and 12 weeks | 4, 8, and 12 weeks
  Difference in the percentage of patients achieving peripheral SBP < 130 mm Hg and/or DBP < 80 mm Hg at t=0 (predose) in patients with uncontrolled hypertension after 4, 8, and 12 weeks of treatment with RTN-001 versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: William CMO, PhD, Study Director — CMO
Locations (3):
- United States (3):
  - Retensiion Clinical Site, Monroe, North Carolina
  - Retension Clinical Site, Charleston, South Carolina
  - Retension Clinical Site, Vienna, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to info@retensionpharmaceuticals.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Retension reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Supporting Information: CSR
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.

REFERENCES:
- See also: Company web site — https://www.retensionpharmaceuticals.com